CLINICAL TRIAL: NCT01579747
Title: Does Ultrasound Improve Procedural Time in the Lateral Popliteal Approach to the Sciatic Nerve in Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nicholas Lam, Associate Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNMLAM_USvsNSobese
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2013-12

CONDITIONS: Postoperative Pain
Keywords: nerve stimulation; ultrasound; sciatic nerve block; popliteal block; obese
MeSH Terms: conditions — Pain, Postoperative; Obesity | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nerve stimulation sciatic nerve block (Placebo Comparator): Time taken to complete a sciatic nerve block via the lateral popliteal approach using nerve stimulation
  Interventions: Procedure: Nerve stimulation
- Ultrasound guided sciatic nerve block (Active Comparator): Time taken to complete a sciatic nerve block via the lateral popliteal approach when using an ultrasound
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Using ultrasound for nerve localization when performing a sciatic nerve block via the lateral popliteal approach
  Arms: Ultrasound guided sciatic nerve block
Procedure: Nerve stimulation — Using nerve stimulation for nerve localization in sciatic nerve blocks via the lateral popliteal approach
  Arms: Nerve stimulation sciatic nerve block

SUMMARY:
Ultrasound have been shown to improve the time needed to locate and block nerves in the non obese population. However, its utility is still unknown in the obese population. Ultrasound is known to produce poorer quality images in the obese population. This study aims to find out if it is a better tool for nerve localization compared to the traditional nerve stimulation technique.

DETAILED DESCRIPTION:
This is a single blinded randomized controlled trial comparing the procedural time for a sciatic nerve block via the lateral popliteal approach using ultrasound compared with nerve stimulation.

24 patients will be randomly selected to determine if the patient will receive their sciatic block using an ultrasound or a nerve stimulation technique.

Patients chosen to receive the ultrasound technique will have their blocks performed by attending regional anesthesiologist who are experts at ultrasound guided sciatic nerve blocks via the lateral popliteal approach.

Patients chosen to receive the nerve stimulation technique will have their blocks performed by attending regional anesthesiologist who are experts at nerve stimulation sciatic nerve blocks via the lateral popliteal approach.

Blinding:

Both the patient and the person assessing the block will be blinded to the group allocation. The highest pain score during the procedure will be obtained by an observer blinded to the group allocation. The time taken for the block, the number of skin punctures and number of passes will be recorded by a person who is not performing the block.

All popliteal blocks will be performed preoperatively by 1 of 4 staff anesthesiologists with substantial expertise in both peripheral nerve localization techniques. Patients will be in the supine position with a bolster below the calf keeping the tibia parallel to the floor. This allows placement of the ultrasound probe in the popliteal region in the ultrasound group. An ultrasound machine and a nerve stimulator will be set up in both groups and the patient will be blinded on the technique used for nerve localization. The ultrasound machine will be turned on and placed perpendicular to the anesthesiologist performing the block on the opposite side of the leg being blocked. The nerve stimulator will be turned on and a grounding lead place on the side of the leg being blocked for both groups. The anesthesiologist performing the block will be given the allocation only after the set up of both systems and just prior to commencement of the block. The patient will be sedated with 2-5mg midazolam and 50-200 ug fentanyl to achieve anxiolysis while maintaining verbal contact. A screen will be set up to prevent the patient or the person assessing the block from seeing the block or the ultrasound screen.

Nerve stimulation group:

Time of block performance starts from first palpation of landmarks to the final injection of local anesthetics. The site of needle insertion was identified and marked (Surgical Skin Marker VX100; Vio Healthcare, Hailsham, East Sussex, UK) as the groove between the biceps femoris and vastus lateralis muscle 10 cm above the top of the patella. (4) A 22G 80mm (SonoPlex Stim Cannula Pajunk Medizintechnologie Germany) insulated needle is inserted with a nerve stimulator set at 1.0mA. The needle is inserted perpendicular to the skin and redirected at a 30 degree angle relative to the horizontal plane. The needle depth is estimated using the midpoint of the thigh and the tangential trajectory of 30 degrees. If plantar flexion is elicited, the nerve stimulator is dialed down to produce a stimulation at 0.4mA or less. If stimulation persists at 0.2mA, the needle is withdrawn until stimulation disappears at 0.2mA but persists below 0.4mA. If dorsiflexion is elicited, the needle is inserted deeper to achieve plantarflexion. Internal rotation of the leg may be help in achieving the angulation.(4) If the needle does not achieve any stimulation, the needle is redirected in 5 degree increments between a 15 to 45 degree trajectory. (5) When the needle is in the correct position, 20 cc of 1.5% mepivacaine is injected in 5 cc increments over 30 seconds. Aspiration for blood is performed before injection and after every 5 cc of injection. Injection is stopped if blood is aspirated or if there is pain on injection. The needle is then repositioned or the block abandoned on the discretion of the anesthesiologist doing the block. However, blood aspiration or pain will be noted.

Ultrasound group

Time of block performance starts from the first antiseptic skin prep on the patient to the final injection of local anesthetics. The lateral and posterior portion of the thigh will be prepped with chlorhexidine. The ultrasound probe is covered with a sterile dressing and placed in the popliteal fossa close to the popliteal crease. The tibial and common peroneal nerve is identified. A long axis slide in the cephalad direction is performed to identify the unity of the tibial and common peroneal nerve into the sciatic nerve. The 28 mm high frequency ultrasound probe is then then moved 2 or more cm cephalad and this is the level of the needle insertion. The 22G 80mm (SonoPlex Stim Cannula Pajunk Medizintechnologie Germany) needle is inserted in-plane from the lateral thigh to approach the sciatic nerve. (6) 20 cc of 1.5% mepivacaine is injected in 5 cc increments over 30 seconds. Aspiration for blood is performed before injection and after every 5 cc of injection. Circumferential spread of local anesthetics around the nerve is sought. The needle is redirected as required to achieve this goal. Injection is stopped if blood is aspirated or if there is pain on injection. The needle is then repositioned or the block abandoned on the discretion of the anesthesiologist doing the block. However, blood aspiration or pain will be noted.

Block Evaluation After the placement of the block, the tibial (bottom of the foot) and common peroneal (top of the foot) will be assessed for motor and sensory loss. Motor loss will be graded as such: 0= no motor strength; 1 = some loss, 2 = full strength. using ice in a PVC glove every 5 minutes for 30 minutes. Sensory loss will be graded as such: 0 = no sensation to ice; 1 = some loss; 2= complete sensation to ice. If the block does not produce complete sensory loss in both distribution within 30 minutes, the block is defined as a failure. It is up to the discretion of the anesthesiologist if he wishes to perform a rescue block or supplement with local field block or to perform a general anesthesia.

Other Evaluation Patients will be followed up in recovery to evaluate if general anesthetic or supplemental local anesthetic by the surgeon is required in the sciatic distribution for surgery.

Patients will be followed up within 72 hours via a telephone interview with regards to signs and symptoms of infection and nerve damage.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Age 18 and above
* BMI >30
* Operations requiring lateral popliteal approach to the sciatic nerve block

Exclusion Criteria:

* Diabetes
* Injection site deformities
* infection at the injection site
* existing peripheral neuropathy
* allergy to LA agents
* Dementia or communication problems
* Inability to understand or discern temperature difference
* Any other contraindication to lower limb peripheral nerve block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Lam, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited in UNMH and outpatient's surgical center
Pre-assignment Details: 1 excluded because not meeting inclusion criteria. Patient lost weight prior to surgery
Groups:
- Nerve Stimulation Sciatic Nerve Block: Sciatic nerve block performed with nerve stimulation
- Ultrasound Guided Sciatic Nerve Block: Sciatic nerve block performed with ultrasound guidance
Period: Overall Study
Arm/Group | Nerve Stimulation Sciatic Nerve Block | Ultrasound Guided Sciatic Nerve Block
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nerve Stimulation Sciatic Nerve Block | Ultrasound Guided Sciatic Nerve Block | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (14.3) | 58.0 (9.4) | 53.65 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Procedural Time
Description: Time taken to complete a sciatic nerve block via the lateral popliteal approach using ultrasound vs nerve stimulation technique
Time Frame: less than 30 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Nerve Stimulation Sciatic Nerve Block | Ultrasound Guided Sciatic Nerve Block
Number analyzed (Participants) | 12 | 12
seconds | 577 (57) | 206 (40)

2. Secondary Outcome: Number of Redirections
Description: Number of needle redirections defined as needle withdrawal followed by advancement as an intentional movement.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: passes
Arm/Group | Nerve Stimulation Sciatic Nerve Block | Ultrasound Guided Sciatic Nerve Block
Number analyzed (Participants) | 12 | 12
passes | 20 [20 to 20] | 3.5 [3 to 4]
Statistical Analysis 1: Comparison: Nerve Stimulation Sciatic Nerve Block vs Ultrasound Guided Sciatic Nerve Block; Normality of distribution was assessed with the Shapiro-Wilk test. For normally-distributed continuous variables, the groups' distributions were described as means and standard deviations (SD). Student's t-test was used to compare groups in these cases with statistically-significant differences summarized using 95% confidence intervals as appropriate. For all comparisons, two-tailed p<0.05 was considered statistically significant; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Nerve Stimulation Sciatic Nerve Block | Ultrasound Guided Sciatic Nerve Block
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
We attempted to minimize performance bias by only involving staff anesthesiologists with years of experience in peripheral nerve blockade using both guidance modalities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No